CLINICAL TRIAL: NCT05819762
Title: Evaluation of ClearLLab LS Screening Panel for the Diagnosis of Hematological Malignancies
Brief Title: Evaluation of ClearLLab LS Screening Panel
Status: Completed | Type: Observational
Sponsor: Beckman Coulter, Inc. (Industry)
Collaborators: Institute of Hematology & Blood Diseases Hospital, China (Other); The First Affiliated Hospital of Soochow University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Tongji Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CHN186
Record Dates: First submitted 2023-03-22; First posted 2023-04-19 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-04

CONDITIONS: Hematologic Malignancy; Hematologic Neoplasms; Hematologic Diseases
MeSH Terms: conditions — Hematologic Neoplasms; Hematologic Diseases | interventions — Flow Cytometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Flow Cytometry — Immunophenotyping of residual clinical samples tested with ClearLLab LS screening panel on a specified Flow Cytometry

SUMMARY:
This is a multi-center study to evaluate the clinical performance of ClearLLab LS screening panel with specimens from subjects for the diagnosis of hematologic malignancies.

DETAILED DESCRIPTION:
This study aims to evaluate the clinical accuracy of ClearLLab LS screening panel in the diagnosis of hematologic malignancies. The residual specimens, which from subjects presenting to the flow cytometry laboratory as part of their standard of care for hematologic diseases work-up, will be tested by ClearLLab LS screening panel. ClearLLab LS screening panel is CE-IVD marked immunophenotyping reagents under the European Union (EU) regulation, and this study is aimed to validate its clinical performance in Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* Residual whole blood, bone marrow, or lymph node tissue samples from subjects with hematologic tumor-related symptoms and/or signs that are clinically recommended for Flow Cytometry Immunophenotyping

Exclusion Criteria:

* Specimens and/or spent samples that are visibly hemolyzed
* Specimens and/or spent samples that are visibly clotted
* Specimens and/or spent samples collected in Ethylene Diamine Tetraacetic Acid (EDTA) anticoagulant older than 24 hours from time of collection
* Specimens and/or spent samples collected in Heparin or Acid Citrate-Dextrose (ACD) anticoagulant older than 48 hours from time of collection
* Samples with insufficient volume to complete the protocol tests
* Samples from subjects with known myeloid malignancies or multiple myeloma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All subjects of any ethnicity, age and racial background will be included
Sampling Method: Probability Sample
Enrollment: 831 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy: sensitivity and specificity | Baseline
  Diagnostic accuracy measured as sensitivity and specificity of ClearLLab LS screening panel in identifying hematological malignancies and non-malignancies compared with the clinical criteria (WHO guidelines)

CONTACTS AND LOCATIONS:
Overall Officials: China Clinical Affaris, Study Director — Beckman Coulter, Inc.
Locations (4):
- China (4):
  - Tongji Hospital, Wuhan, Hubei
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Tianjin

IPD SHARING:
Plan to Share IPD: No